CLINICAL TRIAL: NCT05252598
Title: Mood and Cognitive Effects of Low Doses of Psilocybin Observed in Healthy Subjects ("MELO"): A Blinded, Placebo-Controlled, Dose-Finding Study
Brief Title: Mood and Cognitive Effects of Psilocybin in Healthy Participants
Acronym: MELO
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: The sponsor no longer wishes to pursue the methods outlined in the protocol.
Sponsor: Optimi Health Corporation (Industry)
Collaborators: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB21-1797
Record Dates: First submitted 2022-01-27; First posted 2022-02-23 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Mood Disturbance; Mood Change; Sleep Disturbance; Drug Effect; Psychedelic Experiences; Health, Subjective; Psilocin Toxicity; Psilocybin Toxicity; Psilocybin Causing Adverse Effects in Therapeutic Use; Anxiety
Keywords: Psilocybin; Magic Mushrooms; Microdose; Mood; Sleep; Cognition
MeSH Terms: conditions — Parasomnias; Anxiety Disorders | interventions — Psilocybin; Mezlocillin

STUDY DESIGN:
Intervention Model Description: Participants will be assigned a blister pack containing all the pills for the duration of the study. Each participant will consume 10 capsules each day of the study. The investigational agent will be an encapsulated mushroom powder formulation (derived from Psilocybe cubensis strain) containing varying amounts of psilocybin. The formulation will be altered to ensure each day contains the proposed amount of psilocybin (1, 2, 5, 8, 10mg) or placebo to be tested. Participants and researchers will be blinded to the dose which was consumed on each day of the study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Placebo Arm (Placebo Comparator): 9 placebo pills and 1 non-hallucinogenic Chaga (Inonotus obliquus) mushroom powder capsule to mimic the after-taste of active Psilocybin pills (Psilocybe cubensis)
  Interventions: Drug: Inonotus Obliquus Whole Extract
- 1mg Psilocybin Arm (Experimental): 9 placebo pills and 1 capsule containing encapsulated mushroom powder formulation (derived from Psilocybe cubensis strain) for 1mg of psilocybin
  Interventions: Drug: Psilocybin
- 2mg Psilocybin Arm (Experimental): 8 placebo pills and 2 capsules containing encapsulated mushroom powder formulation (derived from Psilocybe cubensis strain) for 2mg of psilocybin
  Interventions: Drug: Psilocybin
- 5mg Psilocybin Arm (Experimental): 5 placebo pills and 5 capsules containing encapsulated mushroom powder formulation (derived from Psilocybe cubensis strain) for 5mg of psilocybin
  Interventions: Drug: Psilocybin
- 8mg Psilocybin Arm (Experimental): 2 placebo pills and 8 capsules containing encapsulated mushroom powder formulation (derived from Psilocybe cubensis strain) for 8mg of psilocybin
  Interventions: Drug: Psilocybin
- 10mg Psilocybin Arm (Experimental): 0 placebo pills and 10 capsules containing encapsulated mushroom powder formulation (derived from Psilocybe cubensis strain) for 10mg of psilocybin
  Interventions: Drug: Psilocybin

INTERVENTIONS:
Drug: Psilocybin — 1mg encapsulated psilocybin
  Other Names: Melocin
  Arms: 10mg Psilocybin Arm; 1mg Psilocybin Arm; 2mg Psilocybin Arm; 5mg Psilocybin Arm; 8mg Psilocybin Arm
Drug: Inonotus Obliquus Whole Extract — 1mg encapsulated chaga mushroom
  Other Names: Chaga
  Arms: Placebo Arm

SUMMARY:
This study is seeking to find the optimal microdose or low dose of psilocybin (magic mushrooms) that provides general enhancements to mood, memory, sleep, and other measures of general well-being without any hallucinogenic effects.

DETAILED DESCRIPTION:
Psilocybin is a natural psychoactive alkaloid component of more than 200 species of naturally growing mushrooms that can be found throughout the world. Psilocybin use as a ceremonious ritual has been well documented in ancient Aztec and Mesoamerican history. Psilocybin was chemically isolated and synthesized in the 1950s by American scientists, who found that mushroom varieties offered varying ranges of natural psilocybin (from 0.2-1% of dry weight). The psychological benefits of psilocybin are well-documented, as are the safety profile, low toxicity, and significant lack of abuse or overdose potential in comparison to other scheduled and non-scheduled drug, including alcohol. Many clinical studies demonstrate the benefit of psilocybin on feelings of depression, mood, and overall feelings of well-being, particularly at higher doses greater than 25mg. At these doses, hallucinations and psychedelic effects also occur. A growing body of evidence suggests that extremely low doses, or microdoses, may offer similar psychological benefits to individuals without any hallucinogenic effect that may impair daily function. The purpose of this study is to examine an optimal small/microdose of psilocybin, taken orally, that may provide such benefits.

Optimi,is committed to providing MELOCIN, an oral, pharmaceutical grade, but naturally derived, mushroom powder (Psilocybe cubensis), containing a specific dose of psilocybin and a controlled range of other natural compounds and excipients within the formulation. Clinical studies will inform the desired low to very low psilocybin dosing range for specific indications which do not elicit any psychedelic effects but are correlated to specific mood and cognition-related enhancements or improvements in otherwise healthy individuals.

Primary objective: To assess the safety and tolerability of varying low doses and microdoses of Optimi psilocybin-containing mushroom powder in healthy humans.

Secondary objective: To assess the magnitude of effects of varying low doses and microdoses of Optimi psilocybin-containing mushroom powder on general mood, physiological responses, cognitive performance, focus, and feelings of anxiety.

Methodology: Double-blind, randomized, placebo-controlled trial examining effects of six oral doses of MELOCIN, a psilocybin-containing Psilocybe cubensis mushroom powder, with 0 (placebo), 1, 2, 5, 8 and 10mg of psilocybin, administered on six separate test days in a randomized fashion. Participants will be randomized to the order that doses are administered. Study days will be scheduled 6-9 days apart to avoid any carry-over effects of a previous dose. Each study day will require ingestion of 10 capsules, which will be a combination of placebo and Psilocybe cubensis powder containing the prescribed daily dose. On the placebo study day, participants will digest 9 placebo capsules and one Chaga mushroom (non-active, non-hallucinogenic) capsule such that the mushroom after-taste commonly present with hallucinogenic magic mushrooms is mimicked and still present to preserve the blinding of the study dosing regimen.

Participants will be scheduled for 7 total weekly visits (6 dosing days, 1 follow up/close out visit) at the study clinic, each estimated to be 8-9 hours in duration. At each weekly study visit, participants will be continuously monitored and asked to complete cognitive, mood, and other psychological questionnaires and provide minimal blood work at 80-105 mins, 2.5 hrs, 5 hrs, and 7.5hrs post-drug administration in order to monitor the physiological and psychological effects of the dose provided that day. At the follow-up visit, final questionnaires will be completed and qualitative feedback on the experience will be collected

ELIGIBILITY:
Inclusion Criteria:

1. Healthy volunteers
2. Between the age of 18 and 50 years of age
3. Good physical health as determined by medical history, medication history, blood and urinalysis work up
4. Willing to provide informed written consent
5. Able to complete self-assessment questionnaires provided in English
6. Agree to refrain from using any psychoactive drugs, including alcohol, marijuana, or nicotine, at least 24 hours prior to each study visit
7. Agree to refrain from using any non-prescription medication at least 24 hours prior to each study visit

Exclusion Criteria:

1. Unable to complete self-assessment questionnaires in English
2. Reported history of drug abuse or addiction
3. History of any neurological, cardiovascular, or psychiatric disorders or conditions.
4. History, family history in first degree (blood) relatives, or current screening symptoms (as determined by positive mini-international neuropsychiatric interview (MINI) questionnaire) of psychiatric illness (including depression, anxiety disorder, post-partum depression, bipolar disorder, schizophrenia).
5. History of insulin-dependent diabetes mellitus
6. Epilepsy with history of seizures
7. Female participants who are pregnant or nursing
8. Prescribed medications with centrally-active serotonergic or gamma-aminobutyric acid (GABA)-receptor interactions, such as monoamine oxidase inhibitors (MAOI) antidepressants, serotonin-inhibitors (SSRIs) or serotonin-norepinephrine reuptake inhibitors (SNRIs), or neurosteroids
9. Pacemaker or implanted cardiac defibrillator
10. Previous head trauma or concussion history

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-08 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 96 hours post-drug administration
  Collection of data from participants regarding adverse events experience during or after administration of the study drug.
Tolerability of doses with regard to reported hallucinogenic or unpleasant effects (Altered States of Consciousness Scale (5D-ASC), self-reported experience) | Up to 96 hours post-drug administration
  Assessment of hallucinogenic effects or unpleasant side effects assessed using the validated 5D-ASC questionnaire

SECONDARY OUTCOMES:
Assessments of physiological effects of psilocybin capsules | Up to 96 hours post-drug administration
  Use of validated questionnaires to assess drug-effects on mood, sleep, memory, cognition, anxiety and depression

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Taylor, MD/PhD, Principal Investigator — University of Calgary

IPD SHARING:
Plan to Share IPD: No
There is no plan to share data at this time.